CLINICAL TRIAL: NCT05488158
Title: Assessing the Impact of Physician Pain on Motivation to Provide Longitudinal Osteopathic Manipulative Therapy to Patients and Its Correlation to Opioid Prescribing
Brief Title: Assessing the Impact of OMT on Physician Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fort Wayne Medical Education Program (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AOA-Jefferson-1
Record Dates: First submitted 2022-02-23; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MD (Active Comparator): Allopathic physicians in one arm of the study were treated with OMT to alleviate pain and somatic disfunction. The amount of pain they were experiencing before treatment was recorded using a Likert pain scale.
  Interventions: Other: Osteopathic manipulation
- DO (Active Comparator): Osteopathic physicians in one arm of the study were treated with OMT to alleviate pain and somatic disfunction. The amount of pain they were experiencing before treatment was recorded using a Likert pain scale.
  Interventions: Other: Osteopathic manipulation

INTERVENTIONS:
Other: Osteopathic manipulation — Pain and somatic disfunction were treated with osteopathic manipulations as deemed appropriate by a trained DO.

SUMMARY:
Osteopathic Manipulative Therapy/Treatments (OMT) are a non-pharmacologic option for treating patients' pain. As the opioid crisis has developed, the requests for OMT have grown in consequence. This has been associated with a recent focus of opioid addiction and overdose death concerns among physicians and patients. However, the physical toll that OMT takes on the physicians providing the treatments has yet to be robustly investigated. Due to the longitudinal nature of chronic pain, OMT delivery becomes a substantial commitment for the physician offering OMT as an option, especially if the intent is to reduce opioid utilization. Many of the patients treated in our clinic have obesity as a co-morbidity to their chronic pain. The size differential between the patient and provider commonly results in multiple techniques being required to treat the patient's somatic dysfunction, which equates to increased exertion by the provider for each new pain patient. Anecdotal reports from the providers have described a decreased motivation to offer OMT to pain patients due to their own soreness from treating the patients they already have on their panel. Furthermore, the physicians are rarely able to take the time away from their practice during business hours to get their own physical health needs addressed in a timely manner.

This study looked at the participants' pain levels from offering OMT to their patients and their motivation to offer OMT as a non-pharmacological intervention for treating pain. The participants will have protected time built into their schedule where a board certified doctor of osteopathy will treat them every two weeks. Over the study's course, the participants' pain levels and motivation to offer OMT to their patients was assessed. Objective outcome measures came from the participant's patient panel reports. Changes in the number of OMT office visits they provide, the number of systems they treated and the morphine equivalents they prescribed was tracked. The project's hypothesis followed that purposefully attending to the participant's physical health will improve their motivation to offer OMT, reduce their pain and reduce their opioid prescribing.

DETAILED DESCRIPTION:
Physician wellness has become a recent high priority in the medical community. This focus on wellbeing has stemmed from a culture of notoriously high-stress work, long hours, and an increase in publicized physician suicides.8 Many physicians report an increased work burden due to general physician shortages, thus resulting in burn-out. These stressors and associated burn-out are resulting in physicians making the decision to leave the workforce early.9 Mental health initiatives such as Balint groups and peer coaching have been implemented as an effort to combat these concerns.10, 11 As described in greater detail below, very few publications have focused specifically on the physical health considerations of physician wellness.

The Accreditation Council for Graduate Medical Education (ACGME) asks about resident and faculty wellness in their annual programmatic surveys.12 The mechanisms for fulfilling wellness requirements are left to each program to select. This lack of specificity provides programs latitude to meet their own needs, but also doesn't mandate evidence-based approaches. Even the ACGME faculty survey contains questions regarding wellness. ACGME has made the AWARE suite of mobile apps available to residents. The AWARE software is comprised of videos and tools to help residents identify and address burnout or unmitigated stress.13 The Clinical Learning Environment Review (CLER) Pathway to Excellence through the ACGME emphasizes an entire section dedicated to well-being. The well-being pathway in CLER 2.0 calls out "physical and emotional well-being" directly.14 Unfortunately, there are no clear definitions or examples of how a residency program may appropriately meet the required endpoints. The opened-ended nature of this document allows graduate medical education programs to innovate, and address needs specific to each residency program. The well-being section goes on to require programs to demonstrate systems-based approaches in ". . .preventing, eliminating, or mitigating impediments to the well-being of residents, fellows and faculty members".14 The subsections of this pathway requirement only list examples of mental health concerns that could impact residents. There is no direct mention of physical well-being in the document itself.

The primary goal of wellness is to improve the physician's ability to cope with challenging working conditions. To this end, most of the residency programs are focused on mental health.11 Residency programs are working with residents to explore solutions that are most meaningful. The coping strategies developed by residents in training will carry with them into the rest of their careers.15 However, the physical aspects of wellness are noted to be vague and ill-defined. Physicians do report feeling hypocritical when they are encouraging their patients engage in healthy activities, such as exercise, yet are unable to make time for it themselves.16

The inclusion of both mental and physical wellness is imperative according to the Osteopathic principles. Osteopathic approaches to medicine support care for the whole individual. The person's mind, body and soul are understood to be integrated and balanced in a well person.17 It is documented that exercise is known to reduce stress and improve general well-being.18 However, there have been no articles identified that investigated physical health as an independent variable in physician burnout. Delivering osteopathic manipulative treatment as a physician has the potential of creating musculoskeletal discomfort. Physicians have reported soreness and conflicted motivation when scheduling OMT appointments. They want to help their patients and seek to maintain their own well-being simultaneously. Additionally, patients with a larger body habitus may require more exertion to treat. This places physicians in a conflicting mental state, as delivering care could compromise their own sense of comfort and wellness if they offer appropriate patient-centered care.

The role of physician pain in the decision to provide OMT as a modality for patient care necessitates more research. Despite noting that numerous anecdotal reports are made to the faculty of our program each year, we were unable to find published literature specifically addressing this aspect of physician wellness. Numerous publications have addressed physical well-being and patient outcomes.19 For instance, physical pain is a known impediment to regular exercise and lifestyle changes.20 Pain has also been studied extensively for its interference in job performance.21 Due to the physical requirements associated with OMT, physicians who offer OMT services are at a greater risk of soreness. This treatment modality could interfere with the range, scope and frequency of pain management options that are provided to their patient panels. Informal reports have described group sessions where a resident cohort would voluntarily meet outside of traditional work hours to practice OMT on each other as a mechanism to manage individual pain. While valuable as a learning tool, these sessions could be construed as additional patient encounters. It is plausible that these sessions are contributing to physical wear and tear as the residents tend to each other's needs. Additionally, when considering the gatherings as additional patient care encounters, they have the potential to erode work life balance if they feel obligated to treat their peers. Without using social time to get treatment, the physicians wouldn't otherwise have access to care themselves. In this sense, failing to allow for individual treatment could result in canceling patient appointments secondary to physician pain or discomfort. Physicians in these scenarios are continuing to provide treatments on days that would normally be reserved for recuperation.

Anecdotal reports within our family medicine residency program have described feelings of guilt by the physicians who restrict the amount of OMT they perform. They are torn when weighing the option of being physically uncomfortable after providing OMT to a patient versus writing a prescription for an addictive analgesic. We believe that reports of these sentiments have increased for two reasons. First, we are a National Committee for Quality Assurance (NCQA) accredited program.32 This model emphasizes patient-centered care above all. Second, the opioid crisis has our providers seeking as many non-pharmacologic pain management options as possible. When these factors are considered, there are legitimate concerns about how we are to maintain both a patient-centered model and physician physical well-being. Publications on patient centered medical home models have not included the physician in their implementation and delivery paradigms. Furthermore, there are substantially different views on whose well-being takes precedence, patient or physician. For instance, on an airplane the passengers are instructed to secure their own mask before helping others. In healthcare, particularly when OMT is a treatment modality, there is a sense that the doctors must do for others before they do for themselves. In this culture, how then should employers best manage the health of the patient and provider? This study's novelty is rooted in the Osteopathic principles that require the mind, body and soul to be considered holistically when treating patients. Yet these same principles have not been applied to the very physicians who provide longitudinal OMT care to their patients. There are no criteria for what constitutes high frequency or high intensity OMT offerings per week. An iterative and purposeful investigation into the frequency (number of OMT office visits) and intensity of OMT (number of techniques required and number of systems treated) was performed.

Motivation Science: Esteve outlines behavioral impacts of chronic pain as falling into three main categories.42 One such category is the avoidance category, in which patients alter their daily routine to avoid pain or limit their activities to avoid exacerbating their pain. These behavior descriptions match other publications that have focused on the interplay between pain and motivation as well as chronic pain and mental health comorbidities.43 Esteve goes on to discuss "persistence" as a measure of a patient's ability to stick with pain management approaches that foster daily activities. In this way, pain self-management strategies support a patient taking an active role in his or her own care. This approach is like the method for managing other chronic conditions, such as diabetes. Crofford echoes Esteve with the assertion that people will go to greater extents to avoid pain than they would to seek pleasure.44 In these ways, pain can have a clear influence on behavior. It stands to reason those physicians who are constantly sore because of performing OMT routinely on patients would seek to mitigate scheduling those appointments. Furthermore, they may be motivated to prescribe pharmacologic interventions for their patients rather than add additional OMT visits that would exacerbate their own discomfort. In numerous health systems the physician does not play an active role in patient scheduling. As a result, physicians who offer OMT can be over-whelmed with patients in need of longitudinal osteopathic interventions. This lack of scheduling control and its impact on the physicians' well-being has also been anecdotally reported to disincentive offering OMT as a non-pharmacologic chronic pain intervention altogether.

Self-Determination Theory has been used in a variety of settings to explore three different paradigms. The global, contextual, and situational motivations each have precedence over the different experiences a person may face and respond to on a given day. For the purposes of this proposal the focus will be on the contextual paradigm. Based on Vallerand's work Osterlie asserts "The contextual motivation is a motivational disposition towards a particular context, such as work, sports or education."45, 46 With this in mind, the Situational Motivational Scale (SIMS) has been used to assess intrinsic and extrinsic motivation.7 This tool provides an opportunity for assessing correlations between OMT-related patient care, providers' physical wellness, and non-pharmacological pain interventions. These concepts are described in detail below.

The physical toll on the provider (e.g. pain scales or number of systems needing to be treated) has not been compared to the number of systems treated each week, the number of patients receiving OMT, the patient's body habitus (e.g. BMI) or the number of patients provided OMT. These items will be addressed iteratively in the research plan section.

Wellness: Physician wellness is a broad term with numerous programs available.11 Brady's meta-analysis of physician wellness programs looked at 78 publications. Only in 14% of those papers was wellness given an explicit definition. It evaluated both mental and physical health with only a small percentage considering the physician's physical health at all. Lectures on wellness have been incorporated into medical school training globally. Unfortunately, these lectures are didactic in their delivery and the medical students have yet to enter practice. The learners do not know what environment or sub-specialty they will practice in after graduation so the lectures are generalized and lack the specific tools or guidance that the learner will need in the future. The American Medical Society (AMA) has a Steps Forward program designed to assist with wellness, yet its content is also focused on reducing burn out and other mental health related considerations.47 It does not specifically account for the physical considerations of providing patient care. It also describes signs that peers can look out for in a colleague but it does not address the lack of a patient-provider relationship or the use of validated diagnostic tools typically associated with an intervention. This program runs into the same pitfalls that the medical school didactic lectures suffer from in that they are too generic to be a useful skill that students can carry forward into residency. Within residency programs there are a myriad of wellness offerings. For instance, in our program we have a "day of fun" where the cohort goes to an amusement park or other enjoyable activities. These events build an esprit de 'corps but it is an acute intervention and not a purposeful longitudinal program of physical care the physicians need as part of holistic wellness.

Physicians in the Family Medicine Center (FMC) have informally reported that they have attempted to limit the number of osteopathic manipulations performed in a week as a mechanism for protecting their own physical wellness. As mentioned above, the soreness associated with repeated patient manipulations per week reduced the provider's motivation to schedule OMT as frequently within the continuity clinic. Unfortunately, with little control over their scheduling and a workplace culture that puts patients first, physicians usually continue to provide care despite their own discomfort. Providers don't want to "show weakness", disappoint mentors or overload their colleagues. Furthermore, many healthcare organizations have productivity-based metrics. Taking time off work to get care themselves means canceling appointments and disrupting patient care activities. These disruptions may have financial implications, which further demotivates the physicians from ensuring that their health is a high priority. Lastly, admitting they are in pain or physically unable to carry out their duties may influence their workplace relationships.

ELIGIBILITY:
Inclusion Criteria:

* Family Medicine physician residents

Exclusion Criteria:

* Those who did not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Reduction in pain scores | 18 months
  Osteopathic manipulative therapy was employed to treat physician's physical pain as a wellness initiative

CONTACTS AND LOCATIONS:
Locations (1):
- Fort Wayne Medical Education Program, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Dissemination of the aggregate data internally